CLINICAL TRIAL: NCT03898921
Title: Radiofrequency Ablation (RFA) Versus Stereotactic Body Radiotherapy (SBRT) for Small Hepatocellular Carcinoma：A Phase III, Prospective, Randomized, Open, Parallel Controlled Clinical Trial
Brief Title: RFA vs. SBRT for Small HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Clinical Pro., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFA versus SBRT in SYSUCC
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Small Hepatocellular Carcinoma; Radiofrequency Ablation; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): The planned target volume (PTV) was constructed by adding a 5-mm geometric uncertainty margin around the clinical target volume (CTV). The dose-volume constraints used during SBRT planning are fairly standardized: care was taken to ensure that at least 700 cm3 of normal liver parenchyma was exposed to <15 Gy over the course of SBRT, consistent with published recommendation. Radiotherapy dose was prescribed to the isodose surface covering 99.5% of the PTV, typically 75% to 85% of the maximum PTV dose, accepting regional underdosing when necessary to satisfy normal tissue limits.
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)
- Radiofrequency Ablation (RFA) (Active Comparator): Radiofrequency Ablation is carried out under intravenous anesthesia/epidural anesthesia/general anesthesia, with CT or B-ultrasound guidance, through percutaneous or laparoscopic means as far as possible. The ablation range requires complete coverage of the tumor, and has a certain "safe margin". CT/MRI/sonography will be performed 1 month after RFA. If residual tumor was found after treatment, RFA will be carried out again. If there are still residual tumor after two or more RFA treatments, the RFA treatment will be stopped. After the local progression of the tumor, surgical treatment or other treatment methods are considered according to the specific condition.
  Interventions: Procedure: Radiofrequency ablation (RFA)

INTERVENTIONS:
Radiation: stereotactic body radiotherapy (SBRT) — Radiotherapy dose is 36-54 Gy, irradiated in 3 times, every other day, completed within 1 week.
  Arms: Stereotactic Body Radiotherapy (SBRT)
Procedure: Radiofrequency ablation (RFA) — RFA with a safe margin, RFA again if residual,no more than 3 times.
  Arms: Radiofrequency Ablation (RFA)

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the malignant tumors that seriously threaten the health of people. Its morbidity and mortality rank the third and the second among various malignant tumors in China, respectively. Local ablation therapy represented by radiofrequency ablation (RFA) has been recommended as a first-line treatment for small HCC by most international guidelines. Especially for central small HCC, RFA is considered the first-line choice. With the advancement of radiotherapy equipment and the development of precise imaging technology, stereotactic body radiotherapy (SBRT) has become one of the important treatments for liver cancer.Retrospective controlled studies have shown that SBRT is similar to RFA in treating small HCC, and the local control rate may be better than RFA. But there is no high-level evidence to support which treatment is superior. This project aims to conduct a phase III, prospective, randomized, open, parallel controlled clinical study of RFA versus SBRT for small HCC (solitary tumor≤ 5.0 cm). The results will provide potent evidence for the rational and effective treatment of early HCC and the improvement of clinical guidelines for HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the malignant tumors that seriously threaten the health of our people. Its morbidity and mortality rank third and second among various malignant tumors in China, respectively. Liver transplantation, surgical resection, and local ablation are the main curative treatments for early liver cancer. Our team first reported (Ann Surg, 2006) a prospective randomized controlled clinical trial of radiofrequency ablation (RFA) versus surgical resection for small HCC. The results showed that the long-term efficacy of RFA in the treatment of small HCC is similar to surgical resection. Subsequently, Feng et al (J Hepatol, 2012) and Lv et al reported obtained similar research conclusions. At present, local ablation therapy represented by RFA has been recommended as a first-line treatment for small HCC by many international guidelines, especially for small HCC located in central segments.

With the development of radiotherapy equipment and the precision imaging technology, especially the emergence of stereotactic radiotherapy (SBRT), the status of radiotherapy in the treatment of HCC is increasing. SBRT is defined as the use of external irradiation technology, which is divided into several fractions, and the high dose of radiotherapy is accurately delivered into the tumor. As a result, tumor is subjected to high dose and the normal tissue around the tumor is exposed to relatively low dose. Compared with conventional fractionated radiotherapy (CRT), SBRT possessed fewer segmentation times (1 to 6 F), higher fractional doses (5 to 20 Gy), and steeper gradients at the edge of the target region, so it has stronger biological effect. Meanwhile, SBRT can also protect the normal organs better, especially for the radiotherapy of smaller tumors. Multiple clinical studies and meta-analyses have shown that SBRT is superior to traditional CRT in the treatment of HCC, and the side effects are lower in the acute phase. SBRT has become a mainstream technology for HCC, and has been recommended as a routine local treatment for HCC by NCCN guidelines and NCI radiotherapy guidelines.

This project is to conduct a phase III, prospective, randomized, open, parallel controlled clinical study of RFA versus SBRT for small hepatocellular carcinoma (solitary tumor≤ 5.0 cm; initially treated). The primary end point is 3-year overall survival rate. As for secondary end points, we aim to compare 5-year overall survival rate, 1-, 2-, and 3- year progression-free survival (PFS), local control rate, and rate of complications.Stratified analysis will be performed according to tumor size (≤2.0 cm; 2.1-5.0 cm).

Patients enrolled in this clinical trail received either SBRT or RFA depending on the randomization allocation.

As for SBRT group, the treatment follows the protocol below.Immobilization: Patients are immobilized with vacuum bags or styrofoam in the supine position, with the arms raised above the head. 4DCT scanning: Simple breathing training is conducted before simulation, so that the patient can keep breathing quietly and evenly. A plastic box with reflective marker is placed on the patient's anterior abdominal surface where the respiratory amplitude is relatively large, approximately midway between the xiphoid and the umbilicus. The movement of the marker is recorded by an infrared camera, which is converted into breathing curve by computer software. After the breathing curve becomes stable, the CT data of different respiratory phases is collected by 4DCT in axial cine mode. CT scanning region: From 3-4 cm above the diaphragm to the 4th lumbar vertebra. The intravenous contrast is administered during CT scanning and the slice thickness is 3.0 mm. After 4DCT scanning, images are sorted into 10 phases by the software. Each respiratory cycle is divided into 10 respiratory phases, named as CT0% (end-inhalation), CT10%, CT20% (mid-exhalation), CT30%, CT40%, CT50% (end-exhalation), CT60%, CT70% (mid-inhalation), CT80%, CT90%, respectively. Delineation of the target volumes and organs at risk: Gross tumor volume (GTV) and organs at risk (OARs) are contoured on the 20% CT image (mid-exhalation). Then the GTV is registered to the other respiratory phases of 4DCT scan by a physicist using Atlas-based Auto-segmentation (ABAS, Elekta CMS), and the target volumes are modified and confirmed by a radiation oncologist using the standard window/level settings. GTV is defined as the intrahepatic lesion on images. Internal target volume (ITV) is defined as the combined volume of GTVs on 10 respiratory phases. Planning target volume (PTV) is generated by adding a 6-mm margin to the ITV. OARs include liver, kidney, stomach, small intestine, and spinal cord. Normal liver volume is defined as the entire liver minus GTV. Treatment planning: The plan of volumetric modulated arc therapy (VMAT) is designed on the 20% CT image using Monaco TPS (CMS, Elekta) with an optimization algorithm based on a combination of radiobiological and physical cost functions. Monte Carlo algorithm (MC) is performed in the optimization process and a single arc is conducted using FFF mode. Dosimetric evaluation: For PTV, V95% ≥95%, Dmax < 110%, Dmin >90%. For OARs, mean dose to normal liver (MDTNL) < 13 Gy, V15Gy of liver < 35%; Dmean of kidneys <6 Gy, D0.5cc of esophagus < 21 Gy; D0.5cc of stomach < 21 Gy; D0.5cc of small intestine < 21Gy; D0.5cc of colon < 24Gy; D0.5cc of heart < 30 Gy; D0.5cc of ribs < 39 Gy; Dmax of spinal cord < 18 Gy. The planning is evaluated according to the dose volume histogram (DVH) and the dose distribution of each layer. Elekta linear accelerator (Versa HDTM, MLCi2 80 leaves, 0.5 cm MLC) with 6-MV photons are used for treatment. The isocenter of the irradiation field is defined as the geometric center of the PTV, and the prescribed dose is defined as the average dose of PTV. The prescribed dose is maximized while meeting the dosimetric goals. The prescribed dose is 36-54 Gy in 3 fractions administered within 1 week. Plan Validation and Implementation: Dosimetric verification of plan is performed on a Versa HDTM linear accelerator using the three-dimensional semiconductor detection matrix Delta4 (ScandiDos, Uppsala, Sweden) before treatment for each patient. The gamma evaluation criteria were ±3% of 3 Gy and 3 mm of the distance criterion. After the patient's positioning, a 360° scanning is performed using 4D-CBCT prior to each fraction. The automatic bone registration and manual fine-tuning method are used to register the 20% CT image of 4D-CBCT with the planning CT. Then the positioning error data of 6-degree-of-freedom is obtained for online calibration. If the positioning error after calibration is less than 3 mm, the treatment will be delivered.

As for RFA group, contrast-enhanced ultrasonography (CEUS) was carried out for all patients before RFA. RFA was performed with the use of conscious analgesic sedation (intravenous administration of 0.1 mg of fentanyl, 5 mg of droperidol and 0.1 mg of tramadol hydrochloride) and local anesthesia (5 mL of 1% lidocaine) by an anesthesiologist. All procedures were performed percutaneously by one of three ablation experts with 6 to 15 years of experience under real-time ultrasound guidance. The ZW-II RFA system (Dalong South Technical Co., Ltd., Shenzhen, China) was used for ablation. After the single-needle electrode with an exposed tip was deployed to the residual tumor bottom under ultrasound guidance while avoiding critical structures during temporary suspension of respiration. The radiofrequency generator was activated and initiated with 30 W of power. The power was increased by 10 W per minute to 60 W. Tissue impedance was continuously monitored during the ablation, and generator output was adjusted to generator maximum power or until 8 minutes had elapsed. Then, the lesion was rescanned to determine whether the ablative region had covered the whole tumor or a second ablation was required to achieve a satisfactory ablative area. At the end of the procedure, the needle tract was ablated to prevent bleeding and needle track seeding.

This study is expected to complete enrollment in 3 years and to follow up for 3 years.The primary analysis is performed in the intention-to-treat population. Kaplan-Meier curves will be used to describe the patient's recurrence-free survival, and the corresponding statistical data are calculated, such as median progression-free survival (PFS) and bilateral 95% CI. The secondary analysis used a hypothesis test and a two-sided 95% confidence interval(CI) for the first time of the primary recurrence.Kaplan-Meier curves will also be used to describe the patient's disease progression, and calculated the corresponding statistical data, such as the median overall survival(OS) and bilateral 95% CI.Safety assessments will be also performed by comparing adverse events in the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated hepatocellular carcinoma; the diagnostic criteria are based on the "Diagnostic Criteria for Liver Cancer" in the 2017 edition of the "Diagnosis and Treatment of Primary Liver Cancer" by the Department of Health and Medical Administration of the Ministry of Health of China.
2. Single tumor≤5cm in diameter with no vascular invasion, lymph node or distant metastasis.
3. Central type of liver cancer: the shortest distance between tumor and hepatic vein, portal vein, biliary system trunk or first or second branch, or the posterior inferior vena cava of the liver is no more than 1.0cm.
4. No contraindications to RFA and SBRT treatment.
5. KPS≥90.
6. Liver function: Child-Pugh class A; normal liver volume is more than 800cm3.
7. The expected survival of the patient is more than 6 months.
8. The following conditions are met:

   Platelet≥70×109/L; White blood cell≥3.0×109/L; Hemoglobin≥85 g/L; Serum creatinine≤1.5 × upper limit; PT≤3 second extension.
9. Agree to accept postoperative follow-up required by the design of this study.
10. Patients must have the ability to understand and voluntarily sign the informed consent, and must sign an informed consent before starting any specific procedure for the study.

Exclusion Criteria:

1. In combined with severe heart, lung, kidney or other important organ dysfunction, or combined with serious infection or other serious associated diseases (> CTCAE Version 3.0 adverse events of grade 2), that can not tolerate treatment.
2. Patients have a history of other malignancies.
3. Patients have a history of allergic reactions to related drugs.
4. Patients have a history of organ transplantation.
5. Pregnant women, nursing mothers.
6. Patients cannot be performed RFA or SBRT treatment.
7. Patients have other factors that may affect patient enrollment and assessment results.
8. Receiving immunotherapy or targeted therapy.
9. Refuse the follow-up regulations as required by this study protocol and refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-03-10 (Actual); Primary Completion 2021-03-09 (Estimated); Study Completion 2022-03-08 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival rate | From the end of treatment to 3 years
  The percentage of alive individuals after three years of follow-up, with death as the primary endpoint.

SECONDARY OUTCOMES:
5-year overall survival rate | From the end of treatment to 5 years
  The percentage of alive individuals after five years of follow-up, with death as the primary endpoint.
1-, 2-, and 3-year progression-free survival rate | From the end of treatment to 3 years
  After 1, 2, and 3 years of follow-up, the percentage of the alive subjects with no signs of tumor progression. Tumor progression was the end point of follow-up. For patients who suffer unexplained death or other anti-tumor treatment were found before tumor progression, the PFS calculation is up to this point. Determination of tumor progression is based on imaging examination (CT or MRI), and the evaluation criteria refers to the mRECIST criteria.
Local control rate | From the end of treatment to 5 years
  after long-term follow-up, the percentage of the alive subjects with no signs of local tumor progression. The local tumor progression is the end point of follow-up. Definition of local tumor progression is based on imaging examination (CT or MRI), and the evaluation criteria refers to the mRECIST criteria.
Safety profile: incidence of complications | 30 days after the end of treatment
  The safety of the treatment was evaluated by the incidence of complications. Acute complications are defined as the occurrence of adverse events within 30 days of treatment; long-term complications are defined as the occurrence of adverse events 30 days after the end of treatment. Adverse events are defined in accordance with the NCI CTC AE 4.0 standard.

OTHER OUTCOMES:
Tumor response after radiotherapy | From the end of treatment to 2 years
  To assess tumor response using functional magnetic resonance imaging for patients treated with stereotactic body radiotherapy.
Radiation-induced liver injury | From the end of treatment to 1 years
  To assess radiation-induced liver injury using functional magnetic resonance imaging for patients treated with stereotactic body radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: ZHANG YAOJUN, MD., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Feng K, Yan J, Li X, Xia F, Ma K, Wang S, Bie P, Dong J. A randomized controlled trial of radiofrequency ablation and surgical resection in the treatment of small hepatocellular carcinoma. J Hepatol. 2012 Oct;57(4):794-802. doi: 10.1016/j.jhep.2012.05.007. Epub 2012 May 23. PMID 22634125
- [Background] Ng KKC, Chok KSH, Chan ACY, Cheung TT, Wong TCL, Fung JYY, Yuen J, Poon RTP, Fan ST, Lo CM. Randomized clinical trial of hepatic resection versus radiofrequency ablation for early-stage hepatocellular carcinoma. Br J Surg. 2017 Dec;104(13):1775-1784. doi: 10.1002/bjs.10677. Epub 2017 Nov 1. PMID 29091283
- [Background] Lencioni R, Crocetti L. Local-regional treatment of hepatocellular carcinoma. Radiology. 2012 Jan;262(1):43-58. doi: 10.1148/radiol.11110144. PMID 22190656
- [Background] Lau WY, Leung TW, Yu SC, Ho SK. Percutaneous local ablative therapy for hepatocellular carcinoma: a review and look into the future. Ann Surg. 2003 Feb;237(2):171-9. doi: 10.1097/01.SLA.0000048443.71734.BF. PMID 12560774
- [Background] Tateishi R, Shiina S, Teratani T, Obi S, Sato S, Koike Y, Fujishima T, Yoshida H, Kawabe T, Omata M. Percutaneous radiofrequency ablation for hepatocellular carcinoma. An analysis of 1000 cases. Cancer. 2005 Mar 15;103(6):1201-9. doi: 10.1002/cncr.20892. PMID 15690326
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Yoon SM, Lim YS, Park MJ, Kim SY, Cho B, Shim JH, Kim KM, Lee HC, Chung YH, Lee YS, Lee SG, Lee YS, Park JH, Kim JH. Stereotactic body radiation therapy as an alternative treatment for small hepatocellular carcinoma. PLoS One. 2013 Nov 8;8(11):e79854. doi: 10.1371/journal.pone.0079854. eCollection 2013. PMID 24255719
- [Background] Sanuki N, Takeda A, Oku Y, Mizuno T, Aoki Y, Eriguchi T, Iwabuchi S, Kunieda E. Stereotactic body radiotherapy for small hepatocellular carcinoma: a retrospective outcome analysis in 185 patients. Acta Oncol. 2014 Mar;53(3):399-404. doi: 10.3109/0284186X.2013.820342. Epub 2013 Aug 21. PMID 23962244
- [Background] Kimura T, Aikata H, Takahashi S, Takahashi I, Nishibuchi I, Doi Y, Kenjo M, Murakami Y, Honda Y, Kakizawa H, Awai K, Chayama K, Nagata Y. Stereotactic body radiotherapy for patients with small hepatocellular carcinoma ineligible for resection or ablation therapies. Hepatol Res. 2015 Apr;45(4):378-86. doi: 10.1111/hepr.12359. Epub 2014 Jun 16. PMID 24849379